CLINICAL TRIAL: NCT04912817
Title: Pain Rehabilitation Virtual Reality (PR-VR) At-home Program: A Pilot Randomized Controlled Trial to Determine Feasibility and Impact on Pain and Function in Adolescents During and After COVID-19
Brief Title: PR-VR At-home Program During and After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000075493
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pain, Chronic
Keywords: paediatric chronic pain; virtual reality; COVID-19
MeSH Terms: conditions — Chronic Pain; COVID-19

STUDY DESIGN:
Intervention Model Description: A pilot RCT (1:1:1 group allocation) will be used to examine the feasibility of the trial protocol for a definitive trial into the effectiveness of Off-the-shelf VR, Custom VR (Fruity Feet) and Standard Virtual PT (SVPT) in adolescents with chronic pain undergoing functional rehabilitation at home.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Off the Shelf VR (PR-VR program + usual care) (Experimental): * One session per week x 4 weeks; total 4 sessions over 1 month
  * PR-VR program (30 min) + Usual care (30 min SVPT)
  * Total intervention time = 4 hours
  * 10 selected for post-study telephone interview
  Interventions: Other: Off the Shelf VR
- Custom VR (Modified PR-VR program + usual care) (Experimental): * One session per week x 4 weeks; total 4 sessions over 1 month
  * Mod PR-VR program (30 min) + Usual care (30 min SVPT)
  * Total intervention time = 4 hours
  * 10 selected for post-study telephone interview
  Interventions: Other: Custom VR
- Standard Virtual Physiotherapy Treatment (control; usual care), (No Intervention): * One session per week x 4 weeks; total 4 sessions over 1 month
  * Usual care (60 min SVPT)
  * Total intervention time = 4 hours

INTERVENTIONS:
Other: Off the Shelf VR — Operates using Oculus quest VR HMD and uses auditory and visual stimuli during the pain rehabilitation treatment. The Off-the-shelf VR program for Oculus Quest VR features a suite of "off-the shelf" applications that can be tailored by the PT and used with participants including. PR-VR sessions will be 30 minutes in total with approximately 20 minutes in the virtual experience and 10 minutes for set-up, screening, instructions, and rest breaks. The Off-the-shelf VR intervention group will also receive 30 minutes of usual care, and Standard Virtual Physiotherapy Treatment (SVPT) during the same appointment, for a total 1-hour usual care session length.
  Arms: Off the Shelf VR (PR-VR program + usual care)
Other: Custom VR — Operates using Oculus Quest VR HMD with PR-VR software developed with two gaming options: Fruity Feet and Space Burgers 2. Game settings are manipulated by the physiotherapist in session to target specific limb movements and intensity and also motivates participants to cycle using a leg ergometer. Motion sensors on the ergometer track the participants revolutions per minute. For participants in this study arm, a leg ergometer (DeskCycle) will be provided to them during the study phase alongside the Actigraph and Oculus Quest HMD. During the 30min VR portion of the session, 20 minutes will be dedicated to gaming and exercise, and 10 minutes dedicated for set up, tear down, and rest breaks. During the 20 minutes gaming time, a minimum of 15 minutes will be dedicated to Custom VR, with 5 minutes for 'free play' where the participant can opt to try an off-the-shelf VR game.
  Arms: Custom VR (Modified PR-VR program + usual care)

SUMMARY:
Poorly controlled chronic pain in teens can impact quality of life, increase opioid use and is a risk factor for developing chronic pain in adulthood. Currently, there is a shortage of support to help teens manage chronic pain in the community and the support that did exist has been significantly scaled back due to the COVID-19 pandemic. This research study will investigate, based on questionnaires with teens and healthcare providers and interviews with teens, whether pain rehabilitation virtual reality is easy to use and understand, satisfactory to use, and whether it may improve pain, mobility, and function for the teens using the program compared to those doing standard physiotherapy treatment over videoconference.

DETAILED DESCRIPTION:
Chronic pain affects the lives of 1 in 5 - or 2 million - Canadian children and adolescents and has negative impacts on all aspects of health-related quality of life as well as significant economic costs to families and society. The standard of care for pediatric chronic pain management is an interprofessional biopsychosocial treatment approach, a cornerstone of which is physiotherapy (PT) led functional rehabilitation. Furthermore, lack of access to pain clinics and physiotherapy is an ongoing issue which has been exacerbated by the current COVID-19 pandemic; many ambulatory pediatric chronic pain clinics and community-based physiotherapists have halted appointments, with only a few pivoting to virtual service delivery. Providing care virtually is particularly challenging in this field given the physical and hands-on nature pain physical therapy assessment and treatment. These challenges delay treatment and leave vulnerable youth at risk for severe sequelae without the services they require for recovery.

Virtual reality (VR) can help bridge these gaps in care during and beyond COVID-19 by reducing fear associated with movement. A growing body of research has shown the power of immersive VR for reducing anxiety and managing acute pain via distraction in children and adolescents. While there is emerging evidence for the benefit of VR for treating chronic pain in adults, there is minimal research evaluating VR's effectiveness for reducing pain and improving physical function in children and adolescents with chronic pain. Changes to health service delivery due to the COVID- 19 pandemic confirms the crucial need to develop a comprehensive, engaging, and effective approach to home-based chronic pain rehabilitation. The ability of VR to offer patients with chronic pain access to multi-sensory, 3D, immersive therapeutic experiences, has the potential to break the cycle of pain, fear and activity avoidance from a patient's own home.

This pilot randomized controlled trial (RCT) will: (1) Primary Aim: determine the feasibility of implementing an off-the-shelf VR program and custom VR program (i.e., accrual rates, engagement in therapy sessions, retention rates, technical and practical issues, time to set up and conduct PR-VR, treatment acceptability, outcome evaluation, adverse events and participant satisfaction) and; (2) Secondary Aim: evaluate preliminary effectiveness (estimates of magnitude of effect) of VR interventions compared to the usual care condition (standard virtual PT [SVPT]).

ELIGIBILITY:
Inclusion Criteria:

1. able to speak and read English,
2. 12-18 years old,
3. diagnosed with chronic pain,
4. under active care at the interprofessional out-patient Chronic Pain Clinic at SickKids,
5. on stabilized medication/therapy (no new pain medications/therapies for 1 week prior to the initial PT assessment and treatment) according to medical chart,
6. independently mobile and able to safely engage in physical activity,
7. requiring a minimum of 4 treatments (1-hour sessions of virtual PT) typically once per week,
8. able to have access to an Internet-enabled smartphone, computer or tablet at home (typically once per week for 4 weeks) according to self-report for Zoom for Healthcare visits with PT, and
9. willing to have Zoom for Healthcare visits with PT recorded during the study period and, if selected, individual telephone interview with research assistant (RA) audio recorded following the study period.

Exclusion Criteria:

1. visual, auditory or cognitive impairments precluding interaction with the PR-VR intervention and/or control equipment (Internet) as assessed by reviewing the patient's medical chart and consultation with the patient's PT.
2. diagnosis of seizure disorder, history of seizure, or increased risk of seizure.
3. new onset of headaches/migraines, motion sickness, nausea or vomiting or history/symptoms of possible concussion.
4. diagnosis of major, untreated, concurrent psychiatric illness (e.g., depression, anxiety, conversion disorder, PTSD) or personality disorder as assessed by reviewing the patient's medical chart and in consultation by their health care team.
5. currently receiving sedating medications
6. claustrophobia or previous intolerance of virtual reality (e.g. nausea, vomiting, motion sickness, eye strain, false memory formation) as assessed by health care team.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Participant Accrual | 1 year
  PR-VR Recruitment Log has been designed to measure accrual rates (i.e., record data related to the number of eligible adolescents per recruitment day, reasons for ineligibility, and reasons for non-participation)
Participant Engagement | 1 year
  PR-VR Activity Log has been designed to measure participant engagement in the study (i.e., record data related to number of completed sessions as well as independent PT exercise sessions participants self-report completing in between clinician-led sessions)
Participant Retention | 1 year
  PR-VR Activity Log has been designed to measure retention rates (i.e., record data related to reasons for study attrition)
Technical Issues | 1 year
  PR-VR Intervention Log has been designed to record data related to technical and practical issues (occurrence and description) associated with the PR-VR intervention and implementation of the trial protocol, and time to set up and conduct PR-VR as well as any adverse events (e.g. dizziness, nausea) including the date and time the event occurred and the nature of the event.
Safety of PR-VR Program | 1 year
  PR-VR Intervention Log has been designed to record data related to any adverse events (e.g. dizziness, nausea) including the date and time the event occurred and the nature of the event.
Time | 1 year
  PR-VR Intervention Log has been designed to record data related to time to set up
Acceptability/Satisfaction | 1 year
  Measured using the PR-VR Satisfaction Questionnaire completed by adolescent participants and PTs (using adolescent- and PT-specific versions). This questionnaire will collect data on acceptability and perceived utility of PR-VR intervention. Child questionnaire = Scores range from 1-4 (4-pt likert scale), higher scores indicate greater degree of acceptance (better). PT questionnaire = Scores range from 0-4 (5 pt likert scale), each question has different anchors, so better/worse depends on the question
Outcome measure feasibility | 1 year
  Will be measured as the percentage of completed outcome measures at baseline and study completion and will be recorded on the PR-VR Distraction Activity Log

SECONDARY OUTCOMES:
Fear of movement | Collected at baseline (T1) and 4 weeks from baseline (T2)
  Adolescent participants will self-report pain-related fear at T1 and T2 using the Fear of Pain Questionnaire-child (FOPQ-SF). FOPQC-SF scores range from 0 to 40. The total score is the sum of all items on the scale. Cut-off scores for clinical reference groupings are as follows: a score of < 20 indicates Low Fear, 20-25 indicates Moderate Fear and a score of ≥ 26 indicates High Fear.
Pain self-efficacy | Collected at baseline (T1) and 4 weeks from baseline (T2)
  Adolescents will complete the Pain Self-Efficacy Questionnaire (PSEQ), a self-report scale that asks patients to rate their confidence completing an activity/task despite the pain they are experiencing, at T1 and T2. Pain Self-Efficacy Questionnaire (PSEQ) raw scores have a range from 0 - 60. Higher scores indicate greater levels of confidence in dealing with pain.
Pain catastrophizing | Collected at baseline (T1) and 4 weeks from baseline (T2)
  Adolescents will self-report at baseline (T1) and at the endpoint of the study (T2) their tendency to catastrophize about pain during their rehabilitation therapy using the Trait Pain Catastrophizing Scale for Children (PCS-T). PCS raw score is converted to a T-score, where 50 is the mean and 10 is the standard deviation. Higher scores indicate greater pain catastrophizing (worse)
Pain intensity | Collected at baseline (T1), and immediately post- each PT session verbally to the PT, and 4 weeks from baseline (T2)
  Adolescents will self-report their current pain at T1 and T2, as well as pre-, during (10 minutes from the start of their session), and immediately post- each PT session verbally to the PT. Pain will be reported by children using the PROMIS 11-point Numerical Pain Rating Scale (NPRS). NPRS scores range from 0-10 and higher scores indicate greater pain intensity (worse)
Presence/immersiveness | Post- each PT session, through study completion, an average of 1 year
  Adolescents will answer questions regarding how they felt using the virtual reality intervention using the Child Presence Measure post- each PT session. Child presence measure: Scores range from 0-24 with higher scores indicating greater degree of immersion (better)
Exercise intensity | reported verbally to PT Pre-, during (10 minutes from the start of their session), and post- each PT session - through study completion, an average of 1 year
  Self-report modified Borg Scale Rating of Perceived Exertion for Dyspnea and Fatigue (RPE) will be reported verbally to PT pre-, during (10 minutes from the start of their session), and post- each PT session as an indicator of degree of physical strain. Modified Borg RPE scale is Dyspnea and Fatigue are each reported on a scale of 0-10 with higher scores indicating greater dyspnea or fatigue respectively (not necessarily better or worse)
Physical activity levels | 6 months
  An Actigraph (ActiGraph GT9X Link) will be used on participants to record movement during the treatment phase as an objective measure of physical activity levels.
Physical functioning - Mobility | Collected at baseline (T1) and 4 weeks from baseline (T2)
  PROMIS Pediatric Mobility scale will be used to assess participant's perceived difficulty with physical mobility, such as getting out of bed, walking or running. PROMIS Pediatric Mobility (SF), Raw scores are converted to T Scores where 50 is the mean and 10 is the standard deviation. Lower scores indicated greater difficulty with mobility (worse)
Physical functioning - lower extremity | Collected at baseline (T1) and 4 weeks from baseline (T2)
  The Lower Extremity Functional Scale (LEFS) will be used to measure participant's lower extremity function at T1 and T2. LEFS: Scores range from 0-80 with higher scores indicating better functioning (better)
Physical functioning - upper extremity | Collected at baseline (T1) and 4 weeks from baseline (T2)
  Adolescents will self-report upper limb functional impairments using the Upper Extremity Functional Index (UEFI).
Physical functioning - functional disability | Collected at baseline (T1) and 4 weeks from baseline (T2)
  The Functional Disability Inventory (FDI) will be used to assess pain-related disability and functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, RN, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No